CLINICAL TRIAL: NCT05267249
Title: Revascularisation of Autotransplanted Teeth - Retrospective Analysis of a Novel Technique
Brief Title: Revascularisation of Autotransplanted Teeth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ResectTX
Record Dates: First submitted 2022-02-23; First posted 2022-03-04 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-02

CONDITIONS: Endodontic Disease; Pulp Canal Obliteration
Keywords: Autotransplantation, Apicoectomy, Revascularisation
MeSH Terms: conditions — Dental Pulp Diseases | interventions — Transplantation, Autologous; Apicoectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Autotransplantation (Experimental): Autotransplantation and apicoectomy of mature teeth
  Interventions: Procedure: Autotransplantation and Apicoectomy

INTERVENTIONS:
Procedure: Autotransplantation and Apicoectomy — Autotransplantation of a mature teeth with simultaneous extra-oral root-end resectoin

SUMMARY:
Retrospective Analysis of a Study cohort that experienced autotransplantation of mature teeth with simultaneous root end resection

Note: The study was registered on Clinicaltrials.gov after termination of study.

ELIGIBILITY:
Inclusion Criteria:

* Male and female consenting and judicious young people and adults
* Written consent of the participant and, if applicable, of the legal guardian after education
* Planned tooth transplantation with advanced or completed root growth

Exclusion Criteria:

* Contraindications for magnetic resonance imaging (MRI): (pronounced metal restorations, running orthodontics with metal, fixed appliance in the target jaw)
* Current or past antiresorptive therapy with bisphosphonates
* Further anamnestic general or local risk situation, among others: Anti-angiogenic therapy, History of local radiation therapy, severe coagulation disorder, unadjusted diabetes mellitus, malignant diseases
* Acute gingivitis or advanced periodontitis
* Participation in an ongoing drug trial (various drugs may distort the result, such as bisphosphonates, cortisone, chemotherapeutics, angiogenesis inhibitors)
* heavy smokers (> 10 per day)
* Acute or chronic infections (osteomyelitis) at the surgical site
* metabolic diseases (diabetes, hyperparathyroidism, osteomalacia)
* Severe kidney dysfunction, severe liver disease
* Patients with high-dose corticosteroid therapy
* prolonged corticosteroid or radiotherapy in the oral cavity
* autoimmune diseases
* Pregnant or breastfeeding women

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-08-06 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
Survival | 1 year
  Tooth survival

SECONDARY OUTCOMES:
Revascularisation | 1 year
  Occurrence of Revascularisation

CONTACTS AND LOCATIONS:
Overall Officials: Petra Rugani, DDS, Principal Investigator — Medical University of Graz
Locations (1):
- Medical University of Graz, Graz, Styria, Austria

IPD SHARING:
Plan to Share IPD: Undecided
Available upon reasonable request

REFERENCES:
- [Background] Jakse N, Ruckenstuhl M, Rugani P, Kirnbauer B, Sokolowski A, Ebeleseder K. Influence of Extraoral Apicoectomy on Revascularization of an Autotransplanted Tooth: A Case Report. J Endod. 2018 Aug;44(8):1298-1302. doi: 10.1016/j.joen.2018.04.016. Epub 2018 Jun 20. PMID 29935869

DOCUMENTS (1):
  • Study Protocol (2021-07-19): https://cdn.clinicaltrials.gov/large-docs/49/NCT05267249/Prot_000.pdf